CLINICAL TRIAL: NCT05384145
Title: A Type 2 Hybrid Effectiveness-implementation Trial to Evaluate a Population Health Combination Intervention to Meet HIV Testing, Linkage, and Viral Suppression Goals in Coastal Alabama
Brief Title: Implementation Trial to Evaluate a Population Health Combination Intervention to Meet HIV Testing, Linkage, and Viral Suppression Goals in Alabama
Acronym: COAST-AL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Mobile County Health Deparment (Unknown); Alabama Department of Public Health (Unknown)
Responsible Party: Principal Investigator, Aadia Rana, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300009300; 5R01AI169671-03 (NIH)
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: HIV; HIV Linkage to Care; HIV Testing; HIV Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COAST-AL (Other): This combination intervention includes three CDC evidence based interventions: (1) a data-driven approach to direct Community-based HIV testing to areas with high need, (2) Project Connect to expedite linkage to care at time of diagnosis, (3) and a Rapid ART Start program, all in MCHD jurisdictions in Alabama
  Interventions: Other: COAST-AL

INTERVENTIONS:
Other: COAST-AL — This combination intervention includes three CDC evidence based interventions: (1) a data-driven approach to direct Community-based HIV testing to areas with high need, (2) Project Connect to expedite linkage to care at time of diagnosis, (3) and a Rapid ART Start program, all in MCHD jurisdictions in Alabama

SUMMARY:
The purpose of this study is to adapt and evaluate a combination intervention that includes: (1) a data-driven approach to directed community-based HIV testing to areas with high need, (2) Project Connect to expedite linkage to care at time of diagnosis, (3) and a Rapid ART (antiretroviral therapy)Start program, all in Mobile County Health Department (MCHD) jurisdictions in Alabama.

DETAILED DESCRIPTION:
Aim 1. Adapt and integrate COAST-AL using a pre-implementation formative assessment guided by the CFIR. In-depth interviews and clinic observations with community clinic providers, clinic administrators, and MCHD and Alabama Department of Public Health (ADPH) officials will inform targeted Community-based testing, linkage through Project Connect, and Rapid Start into existing work flows (inner setting, process), identify opportunities to use publicly available data to inform testing outreach (outer setting), and explore provider attitudes towards Rapid Start (individuals).

Aim 2. Assess the clinical and implementation effectiveness of COAST-AL in six AL counties served by MCHD. Using RE-AIM, the investigators will evaluate the effects of COAST-AL on clinical and implementation outcomes on progress towards EHE goals. The primary clinical effectiveness outcome is days to viral suppression (VS) for new HIV diagnoses. The primary implementation outcome is the proportion of Zip Code Tabulation Areas with at least 15% of adult population tested for HIV (Reach).

Aim 3. Utilize a community-academic partnership to identify implementation strategies to support maintenance and future dissemination of COAST-AL. Using interviews, concept mapping, and nominal group techniques to inform implementation mapping, the investigators will work collaboratively with local and state health department stakeholders to identify and prioritize implementation strategies to sustain and implement COAST-AL in other health departments across AL and rural EHE(Ending the Epidemic)-focus states.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1 & 3:
* Fit into one of the following categories:

  1) MCHD leadership, 2) ADPH leadership, 3) clinic administrators, 4) outreach testing specialists, 5) linkage coordinators and community health workers, 6) physicians, 7) nurses, 8) counselors all working at HIV care facilities in the six MCHD jurisdiction counties.
* Over the age of 18 years old.

AIM 2: (IDIs)

* Over the age of 13 years old
* Tested for HIV in MCHD jurisdiction from time of COASTAL implementation to 36 months post-implementation start date.

Exclusion Criteria:

* Exclusion criteria include unwillingness or inability to provide informed consent.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to viral suppression | From HIV diagnosis to 1 year
  Effectiveness outcome: Using ADPH EHARS data of all newly diagnosed individuals in MCHD jurisdiction during the study period
Proportion of zctas with >15% population HIV tested | 3 year intervention period
  Implementation outcome: Using commercial lab data sets (Quest/LabCorp) and ADPH data

SECONDARY OUTCOMES:
Proportion linked to care within 30 days | 3 year intervention period
  Effectiveness outcome: Using MCHD FH clinic eHR data
Days from diagnosis to initiation of ART | 3 year intervention period
  Effectiveness outcome: Using MCHD FH clinic eHR data

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No